CLINICAL TRIAL: NCT01355432
Title: Changes in Heart Rate Following Administration of Propofol After Inhalational Induction
Brief Title: Heart Rate Changes With Propofol
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Christopher Lancaster, Attending Anesthesiologist, Nationwide Children's Hospital
Other Study IDs: IRB11-00236
Record Dates: First submitted 2011-05-17; First posted 2011-05-18 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Surgical Patients
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Propofol
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — There is no intervention, this is an observational study.

SUMMARY:
This is a prospective pilot study to quantify the changes in heart rate when propofol is administered after inhalational anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

1. At least 1 year of age or older.
2. Routine (elective) surgical patients with ASA classifications of 1 or 2 (healthy).
3. Patients that are already scheduled to receive inhalational induction followed by IV propofol.

Exclusion Criteria:

1. Premature infants of less than 30 weeks, who are less that 60 weeks post-gestational age at the time of study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgery patients at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in heart rate | Baseline & every 30 secs for 3 mins

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lancaster, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States